CLINICAL TRIAL: NCT01269424
Title: 06-benzylguanine (BG) and Temozolomide (TMZ) Therapy of Glioblastoma Multiforme (GBM) in Patients With MGMT Positive Tumors With Infusion of Autologous P140KMGMT+ Hematopoietic Progenitors to Protect Hematopoiesis
Brief Title: BG & TMZ Therapy of Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanton Gerson MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Stanton Gerson MD, Director, Case Comprehensive Cancer Center, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6307; 8274 (Other: CTEP/NCI); U01CA062502 (NIH)
Record Dates: First submitted 2010-12-31; First posted 2011-01-04 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma Multiforme
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — O(6)-benzylguanine; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): LV gene transfer after concurrent chemo-radiotherapy
  Interventions: Biological: MGMTP140K-encoding retroviral vector; Drug: O6-benzylguanine; Drug: temozolomide; Other: laboratory biomarker analysis; Procedure: autologous hematopoietic stem cell transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: radiation therapy
- Cohort 2 (Active Comparator): LV gene transfer prior to concurrent chemo-radiotherapy
  Interventions: Biological: MGMTP140K-encoding retroviral vector; Drug: O6-benzylguanine; Drug: temozolomide; Other: laboratory biomarker analysis; Procedure: autologous hematopoietic stem cell transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: radiation therapy
- Cohort 3 (Active Comparator): Intra patient dose escalation of TMZ in patients with evidence of P140K marked cells
  Interventions: Biological: MGMTP140K-encoding retroviral vector; Drug: O6-benzylguanine; Drug: temozolomide; Other: laboratory biomarker analysis; Procedure: autologous hematopoietic stem cell transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: MGMTP140K-encoding retroviral vector
Drug: O6-benzylguanine
Drug: temozolomide
Other: laboratory biomarker analysis
Procedure: autologous hematopoietic stem cell transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. O6-benzylguanine may help temozolomide work better by making tumor cells more sensitive to the drug. Giving genetically modified peripheral blood stem cells during or after treatment may prevent side effects caused by chemotherapy.

PURPOSE: This clinical trial studies O6-benzylguanine and temozolomide in combination with genetically modified peripheral blood stem cells in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility of introducing and expressing P140K MGMT cDNA from a lentiviral-based provirus in autologous hematopoietic stem cells harvested from Glioblastoma multiforme (GBM) patients.
* To assess the safety associated with infusion of autologous hematopoietic stem cells transduced ex vivo with a lentiviral vector expressing P140K MGMT in patients with GBM.

Secondary

* To determine whether any patients who receive P140K MGMT-transduced CD34 cells tolerate O6-benzylguanine (BG) and dose-escalated temozolomide (TMZ) without myelosuppression.
* To evaluate the ability to detect P140K-transduced BG and TMZ-resistant hematopoietic cells from the bone marrow and peripheral blood in patients infused with P140K-transduced CD34 progenitors.
* To evaluate the feasibility of in vivo enrichment of P140K-expressing hematopoietic cells by repeated treatments of BG and TMZ at doses that appear therapeutic for GBM.
* To evaluate the efficacy of various types of chemotherapy with or without radiotherapy on conditioning the patient's bone marrow to host the transduced autologous hematopoetic stem cells.
* To evaluate tumor response, progression-free survival, and overall survival.

OUTLINE: Patients are assigned to 1 of 3 treatment cohorts.

* Cohort 1 (LV P140K MGMT gene transfer after concurrent chemoradiotherapy): Patients receive radiotherapy (60cGy in 30 2cGy daily doses) and TMZ 75mg/m2 /daily for 6 weeks, cell infusion at week 7 (T0) followed by BG 120 mg/m2 intravenous infusion over 1h and TMZ 50 mg/m2/day x 5 days, every 28 days (starting on T+28) for 6 cycles.
* Cohort 2 (LV P140K MGMT gene transfer prior to concurrent chemoradiotherapy): Patients receive BG 120mg/m2 intravenous infusion over 1h and TMZ 400 mg/m2 one dose given on day T-2 or T-3 days prior to cell infusion, followed within 72-96 hours by radiotherapy (60cGy in 30 2cGy daily doses) and concurrent BG + TMZ at 50 mg/m2/day x 5 days, every 28 days,starting on T+28 for a total of 7 cycles of BG + TMZ.
* Cohort 3 (intra-patient dose escalation of TMZ in patients with evidence of P140K-marked cells): Dose escalation of TMZ in patients with evidence of P140K marked cells in vivo given as described above for cohort 1 or cohort 2. After completion of radiotherapy, patients will receive BG + TMZ at 50 mg/m2/day x 5 days. Patients not experiencing any grade 3 toxicity will be increased to the next TMZ dose level of 65 mg/m2/day x 5. Subsequent dose escalation without grade 3 toxicity will be 80 mg/m2/day, 100 mg/m2/day, 120mg/m2/day and 140 mg/m2/day x 5. If at subsequent cycles a grade 3 or greater hematologic toxicity occurs, the dose level for the next cycle will be reduced one level.

Blood samples are collected periodically for replication-competent lentivirus detection and other laboratory biomarker studies.

After completion of study therapy, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, newly diagnosed, supratentorial GBM who have undergone gross total tumor resections or near gross total resection (resection of >90% of enhancing tumor demonstrated by MRI) are eligible up to their third post-operative week. Patients with infratentorial disease, multifocal or leptomeningeal disease will be excluded. In general, patients will not have > 1 cm residual measurable or evaluable disease after surgical tumor resection.
* ECOG performance status 0-2 or Karnofsky ≥ 70.
* Patients must have received no myelosuppressive chemotherapy prior to the diagnosis of GBM.
* Life expectancy of at least 12 weeks.
* Adequate hematologic (ANC ≥ 1,000/mm3, platelets ≥ 100,000/mm3, Hgb ≥ 9.5) , hepatic (Bilirubin ≤ 2.0 mg/dl, AST and ALT less than or equal to 3 times upper limit of normal, prothrombin time <1.2 times normal), and renal (Serum creatinine ≤ 2.0 mg/dl or Creatinine Clearance ≥ 60mL/min/1.73 m2 for subjects with serum creatinine levels above institutional normal) . These tests will be repeated within 2 weeks of treatment with BG and TMZ, and must meet the same criteria.
* EKG without evidence of acute cardiac disease.
* Left ventricular ejection fraction (LVEF) ≥ 40
* Post-operative steroids are tapered to ≤ 24 mg decadron/d
* Patients of child-bearing potential must be using single barrier contraception
* Willingness and ability to provide informed consent.
* Patient must have all sutures removed prior to registration
* Patient must be considered to be clinically stable.

Exclusion criteria:

* Medical condition associated with immunosuppression, active infection or medical illness which may jeopardize patient safety.
* HIV seropositivity. This exclusion is included for two reasons. First, there is evidence of decreased marrow reserve in HIV+ patients and antiviral treatment is associated with myelosuppression. Thus, drug treatment designed to be myelosuppressive may be more toxic in this patient population. Second, extensive laboratory culturing of the bone marrow and peripheral blood progenitor cells is required. No preclinical samples which are HIV+ have been evaluated with the gene transfer modality proposed and thus the feasibility and safety of gene transfer and selection in HIV+ samples cannot yet be advocated. Such studies are planned so as to not preclude HIV+ patients in later studies.
* Pregnant or lactating women. There is data to indicate that TMZ is teratogenic and carcinogenic. Thus, its use in pregnant women would confer unnecessary risk to the fetus.
* Patients with symptomatic pulmonary disease and other severe co-morbid conditions
* Patients with cardiac insufficiency and an LVEF of < 40%. History of acute coronary event disease or arrhythmia within 6 months prior to enrollment
* Prior chemotherapy (including gliadel wafers) or hematopoietic cell transplantation.
* Inability to undergo repeated MRI evaluation.
* Prior diagnosis of malignant disease within a three year period with the exception of surgically cured basal cell carcinoma or carcinoma in situ of the cervix
* Mental incapacity or psychiatric illness preventing informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of infusing autologous P140K MGMT-transduced hematopoietic progenitors into patients with GBM | up to 5 years
  Patients will be assessed for clinical symptoms and side-effects - CTCAE v 4.0 - from time of treatment until protocol is stopped due to toxicity, progression, patient choice, or patient election to enroll on new therapeutic option.

SECONDARY OUTCOMES:
Successful transduction rate | up to 4 years
  Quantitate P140K transduced hematopoietic cells from the bone marrow and peripheral blood in patients infused with P140K transduced CD34 progenitors
To evaluate the in vivo enrichment of P140K expressing hematopoietic cells by repeated treatments of BG and TMZ | up to 4 years
  To evaluate the in vivo enrichment of P140K expressing hematopoietic cells by repeated treatments of BG and TMZ
Progression-free | up to 5 years
  Progression-free survival defined as the time interval between the date of initial histological diagnosis and the date of disease progression or death, whichever comes first
Number of patients with radiological progression | up to 5 years
  New tumor or increased tumor size on T1WI + Gd of > 25% as measured by the sum of two perpendicular diameters compared to the smallest measurements ever recorded for the same lesion by the same technique.
Overall Survival | up to 5 years
  From the date of enrollment to death, last contact or last tumor assessment before further anti-tumor therapy, assessed up to 5 years. .

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sloan, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States